CLINICAL TRIAL: NCT05342116
Title: Carbohydrate Rich Drink Reduces Pre-endoscopic Discomfort for Patients Going for Elective Endoscopic Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Ng Wee Khoon, Consultant, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017/00872
Record Dates: First submitted 2022-04-11; First posted 2022-04-22 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Hunger; Depression; Anxiety; Vomiting; Abdominal Pain; Thirst; Fatigue; Lethargy
MeSH Terms: conditions — Depression; Anxiety Disorders; Vomiting; Abdominal Pain; Fatigue; Lethargy | interventions — Water

STUDY DESIGN:
Intervention Model Description: A randomised controlled trial with 3 arms: (1) Fasting 6 hours prior to endoscopy, (2) Allow up to 400ml of water up to 2 hours before endoscopy, (3) Carbohydrate loading with Preload 400ml at least 2-4 hours before endoscopy.
Who Masked: Outcomes Assessor
Masking Description: Endoscopists will be blinded to the patients' assigned arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fasting Arm (No Intervention): Patient will fast at least 6 hours prior to endoscopy
- Water Arm (Active Comparator): Patient will drink 400 ml of water 2 to 4 hours prior to endoscopy
  Interventions: Other: Water
- CHO Arm (Experimental): Patient will drink 400 ml of Preload 2 to 4 hours prior to endoscopy
  Interventions: Other: Nestle Preload

INTERVENTIONS:
Other: Nestle Preload — 1 sachet of Preload (50g) diluted with 400ml of water, to be consumed 2 to 4 hours prior to the endoscopy.
  Arms: CHO Arm
Other: Water — 400ml of water to be consumed 2 to 4 hours prior to the endoscopy.
  Arms: Water Arm

SUMMARY:
The study is a randomised controlled trial that aims to evaluate whether carbohydrate loading pre-endoscopy can improve patients' overall satisfaction and is not associated with negative impact on endoscopic quality or increased complications. A questionnaire will be completed by participants prior to endoscopy.

DETAILED DESCRIPTION:
Currently, the evidence of usage of CHO is mainly for pre-operative patients and has never been evaluated for use in patients before endoscopic procedures which would also require them to fast substantially. Using the same principles of perioperative care, the aim of this a pilot study is to evaluate if Preload usage prior to endoscopic procedures will minimise patient discomfort secondary to fasting with alleviation of preprocedural thirst, hunger and anxiety symptoms. As a result, it may also reduce the urge for patients to drink and ingest prior to endoscopy, which may translate to last minute cancellation of procedures and wastage of precious resources. We believe it will improve overall patient experience and compliance to preprocedural fasting, without significant risks for patients or affecting the quality of endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Planned for elective gastroscopy.
* Able to communicate to give informed consent and complete the questionnaire
* 21 to 80 year old
* ASA physical status I-II

Exclusion Criteria:

* Medications that might impair gastrointestinal motility
* Conditions that may impair gastrointestinal motility, gastroesophageal reflux, pregnancy
* Potential for difficult airway management.
* Diabetic patients.
* American Society of Anesthesiology (ASA) physical status III or more
* Unable to communicate to give informed consent or complete the questionnaire

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluate if Carbohydrate rich drink (CHO) pre-endoscopy improves patients' overall satisfaction. | Questionnaire to be completed 30 to 60 minutes before endoscopy.
  To evaluate if Carbohydrate rich drink pre-endoscopy helps to reduce discomfort experienced by patients during fasting, with lesser thirst, hunger, pain and anxiety, resulting in better overall satisfaction for endoscopic procedures.
  Participants will be asked to complete a Satisfaction Questionnaire prior to the endoscopy.

SECONDARY OUTCOMES:
Evaluate if Carbohydrate rich drink (CHO) pre-endoscopy is safe for patients | Endoscopist Questionnaire will be completed within 60 minutes post endoscopy.
  Most endoscopy centres require patients to fast for 6 to 8 hours prior to endoscopy (fasting arm) or may allow clear fluids up till 2 hours prior to endoscopy (water arm). We aim to evaluate if Carbohydrate rich drink (CHO) has the same safety profile (in terms of risk of aspiration pneumonia and patient discomfort), compared to the conventional fasting arm and water arm.
  Endoscopist performing the gastroscopy will complete an Endoscopist Questionnaire, which will record if there were any periprocedural complications.
Evaluate if Carbohydrate rich drink (CHO) pre-endoscopy affects the quality of gastric preparation | Endoscopist Questionnaire will be completed within 60 minutes post endoscopy.
  Most endoscopy centres require patients to fast for 6 to 8 hours prior to endoscopy (fasting arm) or may allow clear fluids up till 2 hours prior to endoscopy (water arm). We aim to evaluate if Carbohydrate rich drink (CHO) affects the quality of gastric preparation (in terms of good endoscopic views during gastroscopy), compared to the conventional fasting arm and water arm.
  Endoscopist performing the gastroscopy will complete an Endoscopist Questionnaire, which will record if there were good endoscopic views during the gastroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Ng, MBBS, Study Director — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
With the initial pilot study results, we intend to expand it to other endoscopic procedures.

REFERENCES:
- [Background] Gustafsson UO, Hausel J, Thorell A, Ljungqvist O, Soop M, Nygren J; Enhanced Recovery After Surgery Study Group. Adherence to the enhanced recovery after surgery protocol and outcomes after colorectal cancer surgery. Arch Surg. 2011 May;146(5):571-7. doi: 10.1001/archsurg.2010.309. Epub 2011 Jan 17. PMID 21242424
- [Background] Hausel J, Nygren J, Lagerkranser M, Hellstrom PM, Hammarqvist F, Almstrom C, Lindh A, Thorell A, Ljungqvist O. A carbohydrate-rich drink reduces preoperative discomfort in elective surgery patients. Anesth Analg. 2001 Nov;93(5):1344-50. doi: 10.1097/00000539-200111000-00063. PMID 11682427
- [Background] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707
- [Background] Brady M, Kinn S, Stuart P. Preoperative fasting for adults to prevent perioperative complications. Cochrane Database Syst Rev. 2003;(4):CD004423. doi: 10.1002/14651858.CD004423. PMID 14584013
- [Background] Nygren J, Thorell A, Jacobsson H, Larsson S, Schnell PO, Hylen L, Ljungqvist O. Preoperative gastric emptying. Effects of anxiety and oral carbohydrate administration. Ann Surg. 1995 Dec;222(6):728-34. doi: 10.1097/00000658-199512000-00006. PMID 8526579